CLINICAL TRIAL: NCT02625987
Title: Comparison Between Intradermic vs Habitual Skin Closure Technique in Open Appendicectomy.
Brief Title: Appendicectomy Skin Closure Technique: Changing Paradigms (ASC)
Acronym: ASC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: María Valeria Jiménez Baez (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor-Investigator, María Valeria Jiménez Baez, PhD, Coordinación de Investigación en Salud, Mexico
Organization: Coordinación de Investigación en Salud, Mexico (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015-2301-6
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Appendicitis
Keywords: Appendicectomy, wound complications, skin closure
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous intradermic stitch (Experimental): Closure was did with a continuous intradermic stitch.
  Interventions: Procedure: Continuous intradermic stitch
- Separated stitches (Sham Comparator): Like comparator was used a closure with separated stitches.
  Interventions: Procedure: Separated stitches

INTERVENTIONS:
Procedure: Continuous intradermic stitch — Appendectomy wound closure with an intradermic Polyglactina 910 stitch
  Other Names: Subdermic closure with an absorbable suture
  Arms: Continuous intradermic stitch
Procedure: Separated stitches — Appendectomy wound closure with a separated stitches.
  Other Names: Habitual appendectomy wound closure
  Arms: Separated stitches

SUMMARY:
To compare the results associated with two different skin closure techniques in open appendectomy. 200 patients were included after acute appendicitis diagnosis in emergency department. They were grouped randomly into two groups: patients who would receive skin closure with skin closure by an unique absorbable intradermic stitch (Group A) and another that would receive a habitual technique consistent in non absorbable separated stitches (Group B). General characteristics like gender, age, body mass index (IMC), comorbidities and allergies were registered. Days of evolution (DOE) until surgery, use of antibiotics previously, complicated or uncomplicated appendicitis, surgery time and wound complications like skin infection, dehiscence, seroma or abscess were registered in each case too,

DETAILED DESCRIPTION:
Registration number R2015-2301-6 by Local Committee on Ethics in Health Research and Social Security Mexican Institute, Zone 03 General Hospital. The investigators conduct the study at the Hospital General Regional No. 17 in Cancun, Quintana Roo. México. At time in which General Surgery Department determined acute appendicitis diagnosis and prophylaxis antibiotics administered with 3rd generation cephalosporin and Metronidazole, patients receive information about the study and treatment options and informed consent were signed. After this, patients were randomly assigned to one of two study groups. Group A receives a skin closure with a unique absorbable suture intradermal stitch. Group B receives a skin closure with habitual technique, consistent in separated stitch of a non-absorbable suture. The surgical and skin closure techniques were standardized among eight surgeons who participate in the study.

Acute appendicitis diagnosis was established by clinical history, physical exam and laboratory test including blood count, glucose, urea, creatinine, general urinary exam and clothing times. An Alvarado scale >7 points or the surgeon opinion was diagnostic of appendicitis. General information about the patients were recorded like gender, age, body mass index (IMC), comorbidities and allergies were registered. Clinical history information like DOE and previous antibiotics use were registered too.

After explanation of the diagnosis and treatment options, the patients were informed about this study, the objectives, implications, possible outcomes and complications. The patients or legal tutor of the patients refer to understand the possible risk and consequences and if they accept to be included in the study an informed consent was signed.

One hour before skin incision a prophylaxis dose of a 3rd Generation Cephalosporin (Cefotaxime) and Metronidazole were administered. According to a randomized list patients were assigned to one of the two study groups previous to his/her skin incision. The surgical and skin closure technique were standardized and verified by the protocol author previous to the development of any appendectomy by the eight surgeons included in the study.

A Rochy-Davis incision was performed in all cases and aspiration of purulent liquid when required. Stump management with Halsted or Pouchet technique was done. Abdominal cavity was cleaned only with gauze pads, no drain were placed. After aponeurosis closure with Polyglactina 910 #1 continuous point, wound lavage with NaCl 0.9% solution was performed. Dermis was closed with Polyglactina 910 #3-0. In Group A Polyglactina 910 # 3-0 intradermic continuous point was done. In Group B skin closure with Nylon #3-0 separated stitches was achieved.

Liquid diet was ingested 8 hours after surgery and progressed to normal if tolerated. In cases of complicated appendicitis antibiotics were continued four to five days and for uncomplicated appendicitis only by 2 days or until inflammatory systemic response signs were absent. When diet was tolerated and systemic response signs were absent discharge was accomplished.

Surgery incision was evaluated daily until discharge and in extern consult at 7 and 30 days after surgery. In case of group B stitches removal were done at 10 days after surgery.

Days of evolution (DOE) previous to appendicitis diagnose, use of antibiotics previously, complicated or uncomplicated appendicitis, surgery time and wound complications like skin infection, dehiscence, seroma or abscess were registered in each case.

Database was performed and the statistical program SPSS version 22.0 for Mac IOS 7.0 was used to perform statistical data analysis. Complications, surgical and general characteristics were registered and compared between the groups using X2 test. A multivariate analysis was performed for independent variables and the possible association with complications.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Appendicitis diagnosis
* Informed consent signed
* 0-60 age year old
* surgical confirmation of acute appendicitis
* Antibiotic prophylaxis

Exclusion Criteria:

* Appendicitis diagnosis in patients >60 years old
* No antibiotic prophylaxis
* No informed consent signed

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Decrease in wound complications after appendectomy | 1-30 days after surgery
  Complication like wound seroma, infection, dehiscence or abscess would be registered in each one of the two groups and the incidence compared between them to stablish which one is the best option.

SECONDARY OUTCOMES:
Factors associated with appendectomy complications developement | Previous to surgery and during surgery
  General data and surgery data will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Maria Valeria Jimenez Baez, PhD, Study Director — Mexican Social Security Institute

REFERENCES:
- [Derived] Andrade LA, Munoz FY, Baez MV, Collazos SS, de Los Angeles Martinez Ferretiz M, Ruiz B, Montes O, Woolf S, Noriega JG, Aparicio UM, Gonzalez IG. Appendectomy Skin Closure Technique, Randomized Controlled Trial: Changing Paradigms (ASC). World J Surg. 2016 Nov;40(11):2603-2610. doi: 10.1007/s00268-016-3607-x. PMID 27283187